CLINICAL TRIAL: NCT02664233
Title: Connecting Smartphones With Electronic Health Record to Facilitate Behavioral Goal Monitoring in Diabetes Care
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jing Wang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-SN-14-1027; HSC-SN-14-1027 (Other: UTHealth IRB)
Record Dates: First submitted 2015-12-09; First posted 2016-01-26 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Diabetes; Diabetes Mellitus, Type 2; obesity; self-monitoring; goal setting; mobile health; connected health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connected group (Experimental): Patients will use a smart phone and a fitness tracker for self-monitoring of diet and physical activity for 3 months; 3) Smart phones will provide feedback with graphical presentation of self-monitored information to patients; 4) Patient self-monitored information will be integrated into Chronicle Diabetes, so that educators will be able to view this information and give feedback in a follow-up visit.
  Interventions: Behavioral: Mobile and connected health
- Usual diabetes education and care (No Intervention): Participants will receive standard diabetes education and care; each of the recruiting clinics offers diabetes self-management education programs.

INTERVENTIONS:
Behavioral: Mobile and connected health — Patients will use a smart phone and a fitness tracker for self-monitoring of diet and physical activity for 3 months; 3) Smart phones will provide feedback with graphical presentation of self-monitored information to patients; 4) Patient self-monitored information will be integrated into Chronicle Diabetes, so that educators will be able to view this information and give feedback in a follow-up visit.
  Arms: Connected group

SUMMARY:
In order to facilitate the evidence-based goal setting and self-monitoring intervention into the diabetes education practice, the investigator proposes to use Chronicle Diabetes, an electronic system provided available to the American Diabetes Association diabetes education programs, to set patient diet and physical activity goals, and connect patient self-monitoring information collected from smart phones and fitness trackers to Chronicle Diabetes system to facilitate educators' monitoring of patient adherence to their goals.

DETAILED DESCRIPTION:
Specific Aim 1: To develop and test an interface with Chronicle Diabetes to transfer smartphone collected self-monitoring diet and physical activity information from patients to diabetes educators.

Specific Aim 2: To 2a) conduct usability testing and 2b) examine efficacy of this connected interface technology in a 3-month randomized clinical trial in 60 overweight or obese patients with type 2 diabetes in Houston, Texas and Pittsburgh, Pennsylvania.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes
2. Overweight or obese with an BMI > 25
3. Able to read and write English
4. Own a smart phone that is Jawbone compatible

Exclusion Criteria:

1. Currently undergoing current treatment for a severe psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels from baseline to 3 months | baseline and 3 months post enrollment
  Glycemic control will be determined by HbA1c level. HbA1c will be measured using the A1c NOW self check system via a finger stick or extracted from clinical visit data.
Change in weight measures from baseline to 3 months | baseline and 3 months post enrollment
  Participant weight will be measured via a weight scale or via self-report.

SECONDARY OUTCOMES:
Usability of the connected interface technology as indicated by a System Usability Scale | 3 months post enrollment
  The System Usability Scale measures patients' and educators' acceptability, satisfaction, and perceived usefulness of the intervention that is the focus of this study (that is, the connected interface technology within Chronicle Diabetes--Chronicle Diabetes is an electronic diabetes education documentation system to transfer smartphone and wristband collected self-monitoring diet and physical activity information from patients to diabetes educators). Patients and educators are asked to rate each usability item in the scale from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PhD, MPH, RN, Principal Investigator — The University of Texas Health Science Center at Houston, School of Nursing
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Derived] Wang J, Coleman DC, Kanter J, Ummer B, Siminerio L. Connecting Smartphone and Wearable Fitness Tracker Data with a Nationally Used Electronic Health Record System for Diabetes Education to Facilitate Behavioral Goal Monitoring in Diabetes Care: Protocol for a Pragmatic Multi-Site Randomized Trial. JMIR Res Protoc. 2018 Apr 2;7(4):e10009. doi: 10.2196/10009. PMID 29610111